CLINICAL TRIAL: NCT03965247
Title: The Effects of Short-term Lithium Administration on Striatal Reward Processing and Prefrontal Control During Reappraisal in Healthy Volunteers
Brief Title: Lithium Effects on Reward Processing and Reappraisal in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, CatherineHarmer, Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: REC 10/H0605/71
Record Dates: First submitted 2019-04-26; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Lithium; Reward; Caudate; Reappraisal; Prefrontal cortex; Amygdala
MeSH Terms: interventions — Lithium; Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the placebo or lithium group. The two groups were matched in terms of age and gender.
Who Masked: Participant, Investigator
Masking Description: The randomisation schedule was drawn up by an experimenter in the lab who is not involved in the study, and all information was kept in a locked cabinet in the Neurosciences building at the Department of Psychiatry, University of Oxford.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium (Experimental): Increasing amounts of lithium for 11 plus or minus 1 day. Day 1: 400 mg at night Day 2: 600 mg at night Day 3-11: 800 mg at night. The lithium intervention was prepared from 200mg Priadel prolonged release tablets. The intervention was provided in blue and white gelatine capsules to be taken orally.
  Interventions: Drug: Lithium
- Rayotabs (Placebo Comparator): The placebo intervention was 200mg Rayotabs. The intervention was provided in blue and white gelatine capsules to be taken orally - same as the lithium intervention to maintain blinding.
  Interventions: Other: Placebo - Rayotabs

INTERVENTIONS:
Drug: Lithium
  Other Names: Priadel; Lithium carbonate
  Arms: Lithium
Other: Placebo - Rayotabs
  Arms: Rayotabs

SUMMARY:
Bipolar disorder has been associated with blunted activity in regions associated with emotional processing, such as striatal activity during reward anticipation as well as prefrontal activity during reappraisal. Lithium is the most effective treatment in bipolar disorder. Neurochemical and molecular basis of lithium is well known, but how this translates to mood stabilisation is not understood. This study is designed to address how lithium influences reward and emotion regulation processes in humans.

DETAILED DESCRIPTION:
Background:

Bipolar disorder is a relatively common psychiatric disorder for which treatment options are limited. The so-called mood stabiliser, lithium (usually in the form of lithium carbonate) is one of the most commonly used treatments for the disorder, and is effective in treating both acute mania and as a long term maintenance treatment. The investigator's understanding of the pharmacological mechanisms by which lithium exerts its actions is fairly well developed, however there is a lack of understanding of the psychological mechanisms. Within this study the investigators will look at two different types of emotional processing, namely reward anticipation/feedback and emotion regulation, to gain more understanding on how lithium exerts its mood stabilising effects.

Reward processing:

The neural correlates underlying reward anticipation and feedback can be measured with the Monetary Incentive Delay (MID) task, a widely used task for different disorders. Reward anticipation during the MID task has been associated among others, with ventral and dorsal striatum activity. Most critically, bipolar disorder has been associated with blunted reward function of the medial caudate. Reward feedback has been associated with ventral striatum and OFC/vmPFC activity.

Emotion regulation:

One of the most prominent approaches of emotion regulation is reappraisal . Reappraisal has been shown to consistently activate cognitive control regions and to modulate the bilateral amygdala. Insufficient prefrontal control and reduced downregulation of those prefrontal regions of the amygdala while reappraising negative stimuli has been consistently found in bipolar disorder.

Methods:

Using a double-blind, parallel-group design, 37 healthy volunteers (male and female) are randomly allocated to a 11 (+/- 1) day lithium administration or a placebo condition. After the intervention period, all participants undergo fMRI testing with the MID task and the emotional suppression task to assess reward processing and reappraisal of negative stimuli. The participants also complete a visual control task (checkerboard task) and several behavioural tasks and questionnaires. Lithium levels are measured at the end of the intervention period.

Hypothesis:

Based on the literature on bipolar disorder and the mood stabilising effects of Lithium, the investigators expect lithium administration in healthy participants to:

* Increase caudate activity during reward anticipation
* Increase activation of prefrontal control regions as well as increase negative connectivity between those regions and the amygdala during reappraisal

Fidelity check: significant increases in lithium levels in the lithium intervention group compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the study.
* Subject is between 18 and 55 years of age
* Subject has a body mass index (BMI) in the range of 19-30
* Subjects will be physically fit, as assessed by a physical examination by a medical doctor.
* if female and of child bearing age must have a negative pregnancy test for inclusion and must be using two forms of effective contraception.
* Subjects will be fluent English speakers
* Thyroid stimulating hormone and creatinine will be assessed pre-treatment to ensure that these are within healthy range
* non or light smoker < 5 cigarettes per day
* right handed

Exclusion Criteria:

* taking psychotropic medication
* any past or current axis 1 psychiatric disorder on DSM-IV
* Any medical contra-indication (for example, conditions that might alter absorption of lithium or which could impact on the safety of the druk for the volunteer, for example impaired renal function as assessed by creatinine levels or impaired thyroid function as assessed by thyroid stimulating hormone levels)
* Current pregnancy or breastfeeding
* Current or past history of drug or alcohol dependency
* Participant in a psychological or medical study involving the medication within the last 3 months
* Smoker > 5 cigarettes per day
* Dyslexia
* Any contra-indication to MRI scanning, for example chance of metal in the body
* Left-handed

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2012-09-04 (Actual); Study Completion 2012-09-04 (Actual)

PRIMARY OUTCOMES:
brain response to reward anticipation (MID task, Knutson et al. 2001) | Completed during the final day of the intervention period (day 11 (+/- 1) of lithium or placebo treatment).
  Participants are presented with a cue indicating the option to get a reward when responding correctly, no reward when responding correctly, or a cue indicating not to move, while laying in the MR scanner (fMRI study). Group differences in the brain response while anticipating a reward (after reward cue) will be compared to the brain response while not anticipating a reward (after no reward cue). The tested region of brain activation will be restricted to the caudate nucleus and the nucleus accumbens, based on Yip et al. (2015) and Knutson et al. (2001).
Brain response during reappraisal task (Phan et al. 2005) | Completed during the final day of the intervention period (day 11 (+/- 1) of lithium or placebo treatment).
  Participants will perform a reappraisal task (Phan et al. 2005). Trials in which they were asked to either down-regulate negative affect evoked by highly arousing and aversive pictures (e.g., experience naturally) using cognitive reappraisal will be compared to trials where negative affect if maintained. Group differences in brain activation changes during this comparison will be assessed with a specific focus on the prefrontal cortex, as well as on connectivity changes between prefrontal cortex and amygdala during this contrast.

SECONDARY OUTCOMES:
brain activation in response to reward feedback (MID task) | Completed during the final day of the intervention period (day 11 (+/- 1) of lithium or placebo treatment).
  Participants are presented with a cue indicating the option to get a reward when responding correctly, no reward when responding correctly, or a cue indicating not to move, while laying in the MR scanner (fMRI study). After an inter-trial-interfval of 2000-2500ms, a target is presented during which participants need to press a button on reward and no reward trials. If they respond on time it is a hit, otherwise a loss. Group differences in the brain response while receiving feedback on a hit during reward trials will be compared to the brain response while receiving feedback on a loss during reward trials. The tested region of brain activation will be restricted to the caudate nucleus and the nucleus accumbens, based on Yip et al. (2015) and Knutson et al. (2001).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: No
When data was collected, no approval was acquired to share individual participant data. The investigators will make the summary statistics and analyses scripts available.

REFERENCES:
- [Background] Yip SW, Worhunsky PD, Rogers RD, Goodwin GM. Hypoactivation of the ventral and dorsal striatum during reward and loss anticipation in antipsychotic and mood stabilizer-naive bipolar disorder. Neuropsychopharmacology. 2015 Feb;40(3):658-66. doi: 10.1038/npp.2014.215. Epub 2014 Aug 13. PMID 25139065
- [Background] Lahteenvuo M, Tanskanen A, Taipale H, Hoti F, Vattulainen P, Vieta E, Tiihonen J. Real-world Effectiveness of Pharmacologic Treatments for the Prevention of Rehospitalization in a Finnish Nationwide Cohort of Patients With Bipolar Disorder. JAMA Psychiatry. 2018 Apr 1;75(4):347-355. doi: 10.1001/jamapsychiatry.2017.4711. PMID 29490359
- [Background] Knutson B, Fong GW, Adams CM, Varner JL, Hommer D. Dissociation of reward anticipation and outcome with event-related fMRI. Neuroreport. 2001 Dec 4;12(17):3683-7. doi: 10.1097/00001756-200112040-00016. PMID 11726774
- [Background] Oldham S, Murawski C, Fornito A, Youssef G, Yucel M, Lorenzetti V. The anticipation and outcome phases of reward and loss processing: A neuroimaging meta-analysis of the monetary incentive delay task. Hum Brain Mapp. 2018 Aug;39(8):3398-3418. doi: 10.1002/hbm.24184. Epub 2018 Apr 25. PMID 29696725
- [Background] Buhle JT, Silvers JA, Wager TD, Lopez R, Onyemekwu C, Kober H, Weber J, Ochsner KN. Cognitive reappraisal of emotion: a meta-analysis of human neuroimaging studies. Cereb Cortex. 2014 Nov;24(11):2981-90. doi: 10.1093/cercor/bht154. Epub 2013 Jun 13. PMID 23765157
- [Background] Townsend JD, Torrisi SJ, Lieberman MD, Sugar CA, Bookheimer SY, Altshuler LL. Frontal-amygdala connectivity alterations during emotion downregulation in bipolar I disorder. Biol Psychiatry. 2013 Jan 15;73(2):127-35. doi: 10.1016/j.biopsych.2012.06.030. Epub 2012 Aug 1. PMID 22858151
- [Background] Kanske P, Schonfelder S, Forneck J, Wessa M. Impaired regulation of emotion: neural correlates of reappraisal and distraction in bipolar disorder and unaffected relatives. Transl Psychiatry. 2015 Jan 20;5(1):e497. doi: 10.1038/tp.2014.137. PMID 25603413
- [Background] Zhang L, Opmeer EM, van der Meer L, Aleman A, Curcic-Blake B, Ruhe HG. Altered frontal-amygdala effective connectivity during effortful emotion regulation in bipolar disorder. Bipolar Disord. 2018 Jun;20(4):349-358. doi: 10.1111/bdi.12611. Epub 2018 Feb 11. PMID 29430790
- [Background] Hirschowitz J, Kolevzon A, Garakani A. The pharmacological treatment of bipolar disorder: the question of modern advances. Harv Rev Psychiatry. 2010 Sep-Oct;18(5):266-78. doi: 10.3109/10673229.2010.507042. PMID 20825264
- [Background] Phan KL, Fitzgerald DA, Nathan PJ, Moore GJ, Uhde TW, Tancer ME. Neural substrates for voluntary suppression of negative affect: a functional magnetic resonance imaging study. Biol Psychiatry. 2005 Feb 1;57(3):210-9. doi: 10.1016/j.biopsych.2004.10.030. PMID 15691521